CLINICAL TRIAL: NCT04910919
Title: Here's the Buzz: Evaluating Pediatric Post Op Pain and Nausea Following Tonsillectomy Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: competing study started with same participants
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Patti Runyan, Administrative Director, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Buzz Study
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2021-10

CONDITIONS: Tonsillectomy
Keywords: honey; pediatrics; post-operative; pain; nausea; tonsillectomy; complimentary and alternative medicine
MeSH Terms: conditions — Pain; Nausea | interventions — Honey; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): The first 50 participants will receive treatment as usual (alternating weight-based dosing of acetaminophen and ibuprofen with a PRN three-day supply of opioid analgesic).
  Interventions: Other: Standard of Care
- Honey Intervention (Experimental): Participants 51 - 100 will receive the standard of care treatment as usual plus 1 tsp of honey with every dose of acetaminophen.
  Interventions: Dietary Supplement: Honey; Other: Standard of Care

INTERVENTIONS:
Dietary Supplement: Honey — Participants 51 - 100 will receive the standard of care treatment as usual plus 1 tsp of honey with every dose of acetaminophen.
  Arms: Honey Intervention
Other: Standard of Care — The first 50 participants will receive treatment as usual (alternating weight-based dosing of acetaminophen and ibuprofen with a PRN three-day supply of opioid analgesic).

SUMMARY:
Tonsillectomy is one of the most common surgeries performed in the United States, with over half a million performed annually in children younger than 15 years of age. Postoperative pain is one of the most common clinical problems and may lead to poor intake, dehydration, and weight loss. Management of postoperative pain is often challenging and results in additional medical costs due to unplanned emergency room visits. Opioids such as codeine are commonly prescribed for pain control, however in 2013 the Food & Drug Administration issued a black box warning for the use of codeine in post-tonsillectomy pediatric patients. The American Academy of Otolaryngology-Head and Neck Surgery recommends the use of acetaminophen and ibuprofen to successfully manage postoperative pain. With an extended recovery period, often longer than 7 days, alternative measures to reduce postoperative pain are needed. Honey has been proven to possess antibacterial and anti-inflammatory properties. This intervention will evaluate the effect of Tylenol, ibuprofen with honey on children's postoperative pain and nausea following tonsillectomy surgery.

DETAILED DESCRIPTION:
This is a randomized intervention study where 100 pediatric tonsillectomy patients will received standard of care treatment for post-operative pain and randomized by their physician's standing orders on whether or not they include honey for pain management plus the standard of care alternating acetaminophen or Motrin dose (50 patients in the control group and 50 patients in the intervention group).

Patients/ families will be consented for the study during their clinic appointment, by the provider and/ or Registered Nurse (RN) after surgical intervention has been determined as the plan of care or day of surgery if the consent is not present on the EMR by the provider and/ or Holding Room RNs. They will be given a pain catastrophizing scale questionnaire to complete. Patient/ family will be instructed in the use of the medication, pain scale and nausea scale diary by the Holding Room RNs and again with the PACU RNs as they enter they first values before discharge to home. Patients admitted to an inpatient unit are excluded from the study.

The family will be called on post-op Day 1 and Day 4 to answer any questions concerning completing the diary. On Day 5, an image of the diary will be emailed by the family to the PACU for uploading into the secure REDCap database.

Control group families/ patients may call the physician's office postoperatively for pain support and a dose honey may be suggested for post-operative pain. These patients will be grouped into a separately and additional control patients will be enrolled until 50 control patients is achieved.

ELIGIBILITY:
Inclusion Criteria:

* english speaking
* children ages 5-17 years

Exclusion Criteria:

* any child with a genetic syndrome or developmental disability
* allergies to honey
* non-english speaking families

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Numeric value of post-operative pain measured by FACES pain scale | Post-operative day 0 to post-operative day 5.
  The post-operative pain is measured by the self-reported FACES pain scale. The range of scores is from 0-10. 0 (smiling face = no pain) and 10 (crying face) = worst pain ever. This scale is used by patients who are developmentally able, ages 5-9.
Numeric value of post-operative pain measured by Visual Analog Scale (VAS) pain scale | Post-operative day 0 to post-operative day 5.
  The VAS uses a horizontal 10cm line with the extremes of "no pain at all" and "worst pain imaginable". The subject marks on the line their pain rating. Higher points indicate more severe or intense pain. This scale is used by patients who are developmentally able, ages 10-17.
Numeric value of post-operative nausea measured by Baxter Animated Retching Faces (BARF) scale | Post-operative day 0 to post-operative day 5.
  Baxter Animated Retching Faces (BARF) scale has 6 faces with assigned scores ranging from 0 to 10 with a score difference of 2 between each face (a higher score indicates more nausea).

SECONDARY OUTCOMES:
Beliefs and receptiveness of patient families on pain management measured with the catastrophizing scale | Baseline to 6 weeks
  Families will be given a catastrophizing questionnaire to complete to understand their feelings about caring for their child in pain post-operatively. It is a 5 point likert scale that asks participants to select the word that best reflects how strongly they have each questionnaire thought (statement) when their child is in pain, such as 'When my child is in pain, I worry all the time about whether the pain will end', not at all to extremely.

CONTACTS AND LOCATIONS:
Overall Officials: Patti Runyan, DNP, Study Director — Monroe Carell Jr. Children's Hospital at Vanderbilt
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No